CLINICAL TRIAL: NCT02488577
Title: Outcomes Comparison of TAMIS-TME Versus Transanal Minimally Invasive Locoregional Resection for T2 Low Rectal Cancer: an Open Label Study
Brief Title: Outcomes of TAMIS-Total Mesorectal Excision Versus Transanal Loco-regional Excision for T2 Low Rectal Cancer
Acronym: TAMIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Osama Mohammad Ali ElDamshety (Other)
Responsible Party: Sponsor-Investigator, Osama Mohammad Ali ElDamshety, Assistant lecturer of surgical oncology., Mansoura University
Organization: Mansoura University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MISS-TRICKR2
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Low Rectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAMIS TME (Active Comparator): T2 N0 Cases which undergo transanal minimally invasive total mesorectal excision.
  Interventions: Procedure: Transanal minimally invasive total mesorectal excision
- TAMIS-Local (Active Comparator): T2 N0 Cases which will undergo transanal minimally invasive locoregional resection.
  Interventions: Procedure: transanal minimally invasive locoregional resection

INTERVENTIONS:
Procedure: Transanal minimally invasive total mesorectal excision
  Arms: TAMIS TME
Procedure: transanal minimally invasive locoregional resection
  Arms: TAMIS-Local

SUMMARY:
Cases with stage T2 N0 low rectal cancer will undergo either Transanal minimally invasive total mesorectal excision or transanal minimally invasive locoregional resection.

ELIGIBILITY:
Inclusion Criteria:

* T2 N0 low rectal cancer

Exclusion Criteria:

* patients unfit for laparoscopic resection
* Unwilling to share in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Overall percent of postoperative complications. | 30 days
  the over all percentage of Postoperative complications concerning Pelvis abscess, anastomosis disruption, bleeding, Fistula and continence function.

SECONDARY OUTCOMES:
Hospital stay | 30 days
  Number of Days starting from the admission till discharge
Recurrence. | 2 years
  number of local and distant recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Kotb, M.D., PhD., Study Director — Professor of surgical oncology Mansoura university; Osama Eldamshety, PhD, Principal Investigator — surgical oncology Mansoura university; Adel Fathi, M.D., Principal Investigator — surgical oncology Mansoura university